CLINICAL TRIAL: NCT00148746
Title: Standardized Time- and Score-oriented Treatment of Moderate and Severe Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DERMA_AD_001
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Moderate to Severe Atopic Dermatitis
Keywords: atopic dermatitis, atopy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus; Tacrolimus; Prednisolone; Cyclosporins; prednicarbate

INTERVENTIONS:
Drug: Pimecrolimus
Drug: Tacrolimus
Drug: Prednisolone
Drug: Ciclosporin A
Drug: Dermatop

SUMMARY:
The study was designed to test the hypothesis whether a standardized, time-and score-oriented treatment following a strict evidence based algorithm is equally effective to a standard treatment regimen for moderate to severe atopic dermatitis.

Study Type: Mono-centre study, patients are blinded, physicians are randomized to either treat study- or controll group

Eligible are patients age 2 years or older with SCORAD >= 20 Duration: 12 Months, study visits every 4 weeks.

Primary endpoint is Difference between Baseline SCORAD and mean SCORAD under treatment.

Secundary endpoints are quality of life, safety and economic burden in both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe atopic dermatitis (SCORAD 20 or more) fulfilling the diagnostic criteria by Raika and Hanifin

Exclusion Criteria:

* Pregnancy
* Nursing
* Women in childbearing age without contraception
* Drug - and or alcohol abuse
* Gene defects that are associated with increased light sensibility, e.g. Xeroderma pigmentosum, Cockayne Syndrome, Bloom Syndrome

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-05; Primary Completion 2006-09 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jochen M Schmitt, MD, MPH, Study Director — Dpt. of Dermatology, Medical Faculty, Technical University Dresden, Germany
Locations (1):
- Department of Dermatology, TU Dresden, Dresden, Germany

REFERENCES:
- [Derived] Schmitt J, Meurer M, Schwanebeck U, Grahlert X, Schakel K. Treatment following an evidence-based algorithm versus individualised symptom-oriented treatment for atopic eczema. A randomised controlled trial. Dermatology. 2008;217(4):299-308. doi: 10.1159/000151355. Epub 2008 Aug 15. PMID 18703875